CLINICAL TRIAL: NCT06933524
Title: An Open-Label, Multicenter, Phase 1 Clinical Trial to Evaluate the Safety and Tolerability of ATB-320 in Patients With Progressive or Metastatic Solid Tumors
Brief Title: Evaluation of Safety and Tolerability of ATB-320 in Participants With Progressive or Metastatic Solid Tumors
Acronym: ATB-320-001A
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Autotelicbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATB-320-001A
Record Dates: First submitted 2025-04-04; First posted 2025-04-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATB-320 (Experimental): Participants will receive ATB-320 in cycles. One cycle will consist of 4 weeks (28 days). The study will start with Cohort 1 and the progression to the next cohort will depend on the occurrence of dose limiting toxicity (DLT).
  The dosage regimen of the investigational product is as follows:
  Cohort 1: 1.0 mg/kg Cohort 2: 2.0 mg/kg Cohort 3: 4.0 mg/kg Cohort 4: 8.0 mg/kg
  Interventions: Drug: ATB-320

INTERVENTIONS:
Drug: ATB-320 — IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ATB-320 in patients with progressive or metastatic solid tumors

DETAILED DESCRIPTION:
1. Primary objective: to evaluate the maximum tolerable dose (MTD), recommended phase 2 dose (RP2D), and dose limiting toxicities (DLTs) of ATB-320 in patients with progressive or metastatic solid tumors.
2. Secondary objective: to evaluate safety and tolerability of ATB-320 in patients with progressive or metastatic solid tumors.
3. Exploratory objective: to evaluate pharmacokinetics, pharmacodynamics, and efficacy of ATB-320 in patients with progressive or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years or older) at the time of screening
2. Histologically confirmed solid tumor
3. Participants must have failed standard therapy or cannot tolerate standard therapy.
4. Participants must be able to provide tissue samples, either stored at the institution or obtained from a biopsy performed prior to administration of the investigational product, and have tumor that can be safely biopsied throughout the study.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
6. Life expectancy of ≥ 12 weeks

Exclusion Criteria:

1. Has received chemotherapy within 21 days prior to the first planned dose of the investigational product, or if less than 5 times the half-life of the chemotherapeutic has passed (whichever is shorter)
2. Has received immunotherapy within 2 weeks of the first planned dose of investigational product
3. Major surgery within 4 weeks prior to the first planned dose of the investigational product
4. Previous malignant tumors, other than the target indication to be investigated in this study, within 3 years prior to screening (participants with locally malignant tumors such as basal cell carcinoma/squamous cell carcinoma of the skin, carcinoma in situ (cervix, breast), thyroid papillary carcinoma that have undergone potentially curative therapy are eligible to participate in the study.
5. Current enrollment in any other clinical trial or has received another investigational product or medical device treatment within 28 days of first planned dose (participants who are undergoing safety follow-up phase of a clinical trial may participate if more than 28 days have passed since the last dose of the previous investigational product)
6. Has received prior radiotherapy within 2 weeks of the first planned dose. Participants who have received palliative radiotherapy for non-central nervous system (CNS) disease within 2 weeks of first planned dose are allowed to participate after 1-week washout (participants must have recovered from any radiation-related toxicities, not require corticosteroid treatment, and without radiation pneumonitis)
7. History of hypersensitivity to the active ingredients or excipients of the investigational product or other drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | First dose to Cycle 1 Day 28 (each cycle is 28 days)
  Occurrence of dose limiting toxicity (DLT) will be assessed for the DLT Analysis Set for each cohort until Cycle 1 Day 28 (C1D28) and will be discussed by the Data Monitoring Committee (DMC).
Maximum Tolerated Dose (MTD) | At the end of Cycle 1 (each cycle is 28 days)
  The highest dose (cohort) at which no more than one out of three to six participants in a cohort experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Safety | At the end of each cycle (each cycle is 28 days) and up to 14 days from the last dose of ATB-320
  Number of participants with AE, with abnormal physical examination findings, abnormal vital signs, abnormal ECG readings, abnormal clinical laboratory tests results

IPD SHARING:
Plan to Share IPD: No